CLINICAL TRIAL: NCT05348031
Title: Multimodal Analysis of Structural Voice Disorders Based on Speech and Stroboscopic Laryngoscope Video
Status: Not yet recruiting | Type: Observational
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Collaborators: Duke Kunshan University (Other)
Responsible Party: Sponsor
Other Study IDs: SYSEC-KY-KS-2022-040
Record Dates: First submitted 2022-04-19; First posted 2022-04-27 (Actual); Last update posted 2022-04-27 (Actual); Status verified 2022-03

CONDITIONS: Voice Disorders
Keywords: deep learning; multimodality; structural voice disorders; stroboscopic laryngoscope video; Speech
MeSH Terms: conditions — Voice Disorders; Speech

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study intends to collect clinical data such as strobary laryngoscope images and vowel audio data of patients with structural voice disorders and healthy individuals, and to establish a multimodal voice disorder diagnosis system model by using deep learning algorithms. Multi-classification of diseases that cause voice disorders can be applied to patients with voice disorders but undiagnosed in clinical practice, thereby assisting clinicians in diagnosing diseases and reducing misdiagnosis and missed diagnosis. In addition, some patients with voice disorders can be managed remotely through the audio diagnosis model, and better follow-up and treatment suggestions can be given to them. Remote voice therapy can alleviate the current situation of the shortage of speech therapists in remote areas of our country, and increase the number of patients who need voice therapy. opportunity. Remote voice therapy is more cost-effective, more flexible in time, and more cost-effective.

DETAILED DESCRIPTION:
1. Detection and Classification of Acoustic Lesions Based on Speech Deep Learning
2. Detection and Classification of Acoustic Lesions Based on Deep Learning of Images
3. Detection and Classification of Acoustic Lesions Based on Deep Learning Based on Multimodality

ELIGIBILITY:
Inclusion Criteria:

Laryngeal cancer, laryngeal precancerous lesions, benign laryngeal lesions with voice disorders, healthy people without throat diseases

Exclusion Criteria:

1. A history of laryngeal surgery
2. Patients with voice disorders caused by various causes except laryngeal cancer, laryngeal precancerous lesions, and benign laryngeal lesions
3. The audio quality is not clear, the stroboscopic laryngoscope does not clearly display the anatomical area related to the glottis, and it is underexposed and blocked;

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: In this study, 490 patients with voice disorders (including laryngeal cancer, laryngeal precancerous lesions, and benign laryngeal lesions) and 50 healthy people were collected from stroboscopic laryngoscopy videos and vowel audio recordings. Gender, course of disease, VHI and other clinical data.
Sampling Method: Non-Probability Sample
Enrollment: 1 (Estimated)
Dates: Start 2022-05-06 (Estimated); Primary Completion 2025-12-30 (Estimated); Study Completion 2027-02-20 (Estimated)

PRIMARY OUTCOMES:
Machine deep learning classifies vocie disorders | May 6,2022-December 30,2023
  Accuracy
Machine deep learning classifies vocie disorders witn multimodality | January 1,2024-December 30,2024
  precision
Machine deep learning classifies pathological voice change in Laryngeal Cancer | January 1,2024-December 30,2025
  precision

SECONDARY OUTCOMES:
Machine deep learning classifies vocie disorders witn multimodality | January 1,2024-December 30,2025
  recall

CONTACTS AND LOCATIONS:
Overall Officials: YueXin Cai, Study Chair — Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Martínez, David, Lleida Eduardo, Ortega Alfonso,Miguel Antonio, Villalba Jesús. Voice pathology detection on the Saarbrücken voice database with calibration and fusion of scores using multifocal toolkit. Advances in Speech and Language Technologies for Iberian Languages. Springer, Berlin, Heidelberg, 2012. 99-109
- [Background] Hegde S, Shetty S, Rai S, Dodderi T. A Survey on Machine Learning Approaches for Automatic Detection of Voice Disorders. J Voice. 2019 Nov;33(6):947.e11-947.e33. doi: 10.1016/j.jvoice.2018.07.014. Epub 2018 Oct 11. PMID 30316551
- [Background] Al-Nasheri A, Muhammad G, Alsulaiman M, Ali Z. Investigation of Voice Pathology Detection and Classification on Different Frequency Regions Using Correlation Functions. J Voice. 2017 Jan;31(1):3-15. doi: 10.1016/j.jvoice.2016.01.014. Epub 2016 Mar 15. PMID 26992554
- [Background] .Chuang, ZY,YuXT,Chen JY, Hsu YT,Xu ZZ,Wang CT,Lin FC,Fang SH. DNN-based approach to detect and classify pathological voice. In Proceedings of the 2018 IEEE International Conference on Big Data (Big Data), Seattle, WA, USA, 10-13 December 2018
- [Background] Fang SH, Tsao Y, Hsiao MJ, Chen JY, Lai YH, Lin FC, Wang CT. Detection of Pathological Voice Using Cepstrum Vectors: A Deep Learning Approach. J Voice. 2019 Sep;33(5):634-641. doi: 10.1016/j.jvoice.2018.02.003. Epub 2018 Mar 19. PMID 29567049
- [Background] Bethani Gty As H , Suwandi, Anggraini C D . Classification System Vocal Cords Disease Using Digital Image Processing.The 2019 IEEE International Conference on industry 4.0,Artifical Intelligence,and Communications Technology.2019.129-132
- [Background] Unger J, Lohscheller J, Reiter M, Eder K, Betz CS, Schuster M. A noninvasive procedure for early-stage discrimination of malignant and precancerous vocal fold lesions based on laryngeal dynamics analysis. Cancer Res. 2015 Jan 1;75(1):31-9. doi: 10.1158/0008-5472.CAN-14-1458. Epub 2014 Nov 4. PMID 25371410
- [Background] Xiong H, Lin P, Yu JG, Ye J, Xiao L, Tao Y, Jiang Z, Lin W, Liu M, Xu J, Hu W, Lu Y, Liu H, Li Y, Zheng Y, Yang H. Computer-aided diagnosis of laryngeal cancer via deep learning based on laryngoscopic images. EBioMedicine. 2019 Oct;48:92-99. doi: 10.1016/j.ebiom.2019.08.075. Epub 2019 Oct 5. PMID 31594753
- [Background] Kim H, Jeon J, Han YJ, Joo Y, Lee J, Lee S, Im S. Convolutional Neural Network Classifies Pathological Voice Change in Laryngeal Cancer with High Accuracy. J Clin Med. 2020 Oct 25;9(11):3415. doi: 10.3390/jcm9113415. PMID 33113785
- [Background] Godino-Llorente JI, Gomez-Vilda P. Automatic detection of voice impairments by means of short-term cepstral parameters and neural network based detectors. IEEE Trans Biomed Eng. 2004 Feb;51(2):380-4. doi: 10.1109/TBME.2003.820386. PMID 14765711
- [Background] Ren J, Jing X, Wang J, Ren X, Xu Y, Yang Q, Ma L, Sun Y, Xu W, Yang N, Zou J, Zheng Y, Chen M, Gan W, Xiang T, An J, Liu R, Lv C, Lin K, Zheng X, Lou F, Rao Y, Yang H, Liu K, Liu G, Lu T, Zheng X, Zhao Y. Automatic Recognition of Laryngoscopic Images Using a Deep-Learning Technique. Laryngoscope. 2020 Nov;130(11):E686-E693. doi: 10.1002/lary.28539. Epub 2020 Feb 18. PMID 32068890
- [Result] Bainbridge KE, Roy N, Losonczy KG, Hoffman HJ, Cohen SM. Voice disorders and associated risk markers among young adults in the United States. Laryngoscope. 2017 Sep;127(9):2093-2099. doi: 10.1002/lary.26465. Epub 2016 Dec 23. PMID 28008619